CLINICAL TRIAL: NCT03244579
Title: Studying the Effectiveness of Carbohydrate Counting and Dietary Approach to Stop Hypertension Dietary Intervention on Glycemic Control and Maternal and Newborn Health Outcomes Among Jordanian Pregnant Women With Gestational Diabetes
Brief Title: Carbohydrate Counting and DASH Intervention and Pregnancy Outcomes Among Women With Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Sabika Salem Allehdan, Principal Investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2017-07-31; First posted 2017-08-09 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Gestational Diabetes Mellitus With Baby Delivered
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary intervention CHO counting (Experimental): Carbohydrate counting diet will be prepared according to Kulkarni, (2005). Tailored diet plans according to patient's food preference, physical activity level and appropriate insulin: Carbohydrates ratio will be prescribed for each participants. Diets were based on each participants's recommended intakes of energy, protein (15-25%), fat (30-40%) and carbohydrate (40-50%) (Thomas and Gutierrez, 2005; Kleinwechter et al., 2014). Energy requirement will be determined in the participants' pre-pregnancy weight with adding the extra requirement (450 kcal) due to pregnancy. The carbohydrate counts will be distributed into three main meals and 3 snacks.
  Interventions: Behavioral: Dietary Intervention
- Dietary intervention CHO Counting & DASH (Experimental): The recommended intakes of energy, protein (15-25%), fat (30-40%) and carbohydrate (40-50%) will be similar to that in carbohydrate counting diet which mentioned above. DASH diet food choices will be inserted in the diet of the participants assigned for the combined diet of DASH and carbohydrate counting. The emphasis will be more on the fruits and vegetables group (>8 servings/day), whole grains (at least half of the amount of the total servings of cereals; 6-8 servings/day), fat free dairy products (2-3 servings/day), lean meat and plant proteins (0-2 servings/day) and nuts (5-7 servings/week). From the fat group olive oil will represent the main type of fat (20-25% of total fat %). Adequate intake of sodium (2000mg) will be applied into participants' diet.
  Interventions: Behavioral: Dietary Intervention
- General Dietary guidlines (No Intervention): the general dietary advice and diet that will be prescribed by hospital for participants

INTERVENTIONS:
Behavioral: Dietary Intervention — Adjusting the quantity and quality of food intake to improve glycemic control, maternal and newborn health outcomes of women with gestational diabetes.
  Other Names: diet therpy
  Arms: Dietary intervention CHO Counting & DASH; Dietary intervention CHO counting

SUMMARY:
Study is an interventional clinical trial. Pregnant women (aged 25-40 years) diagnosed with GDM (by a 75-g oral glucose tolerance test at 24-28 weeks' gestation) will be recruited conveniently from Obstetrics and Gynecology clinic at the Jordan University Hospital and National Center for Diabetes, Endocrinology and Genetics, Amman, Jordan. A sample of 180 pregnant women with GDM (60 women who do not use insulin and hypoglycemia medications, 60 women who are treated with metformin, 60 women who are treated with insulin), who will meet the inclusion criteria and will be agreed to participate will be centrally randomized to follow carbohydrate counting dietary intervention, carbohydrate counting and DASH dietary intervention, and control dietary intervention.

DETAILED DESCRIPTION:
The main objective of this study is to compare the effect of carbohydrate counting, carbohydrate counting and DASH diet dietary interventions and a general dietary intervention on glycemic control, maternal and neonatal outcomes among Jordanian pregnant women with GDM. Eligibility criteria to be enrolled in the study will be being Jordanian pregnant women with GDM at 24 -28 gestational weeks, aged between 25 to 40 with no-personal history of type 1 or 2 diabetes, or impaired fasting glucose, or chronic diseases and singleton gestation. DASH diet; and the third group will follow the diet prescribed by the hospital for GDM. The duration of intervention will extend from 24-28 gestational weeks until delivery, which will be usually 12-14 weeks later. The glycemic controls outcomes are testing fasting blood glucose, HbA1C, insulin and fructosamine at baseline and at end of intervention for three dietary interventions. While maternal outcomes are total maternal weight gain (kg), need for emergency caesarean section, the presence or absence of pregnancy-induced hypertension and preeclampsia. The new born birth weight, length and head circumference, the presence or absence of hypoglycemia and shoulder dystocia are the newborn outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Jordanian pregnant women with GDM at 24 -28 gestational weeks.
* Aged 25-40 with no-personal history of type 1 or 2 diabetes, or impaired fasting glucose (Koivusalo et al., 2016).
* Singleton gestation (Louie et al., 2011).
* Absence of chronic diseases such as hypertension, hepatic and kidney disease and cancer, and psychiatric disorder (Ma et al., 2014).
* Absence of the use of medication that influences glucose metabolism, such as continuous therapy with oral corticosteroids (Koivusalo et al., 2016)
* Pregnant women who do not have special dietary requirements (Louie et al., 2011).

Nonsmoker or nonalcoholic drinker during pregnancy (Louie et al., 2011) Well educated and well cooperative, more than 10 years of formal schooling (Ma et al., 2014).

Exclusion Criteria:

* Non- Jordanian pregnant women or Jordanian pregnant women with GDM at <24 or >28 gestational weeks.
* Aged > 40 years with multiple gestation and suspected over-diabetes (Koivusalo et al., 2016).
* Multiple gestations (Louie et al., 2011).
* Presence of chronic diseases, severe psychiatric disorder. Women with the risk factors for placental insufficiency, or history of preeclampsia (Ma et al., 2014; Koivusalo et al., 2016).
* Presence of the use of medication that influences glucose metabolism, such as continuous therapy with oral corticosteroids (Koivusalo et al., 2016)
* Pregnant women who have special dietary requirements (Louie et al., 2011).
* Who smoked or consumed alcohol during pregnancy (Louie et al., 2011)
* Less than 10 years of formal schooling or previous intensive nutrition education or intervention for diabetes (Ma et al., 2014).

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2019-08-20 (Estimated); Study Completion 2019-10-20 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | one year
  Fasting blood glucose in mg/dL at 24 -28 weeks of gestation (baseline) and at 36-37) weeks of gestation(endline) of intervention.

SECONDARY OUTCOMES:
Hemoglobin A1c level | one year
  Hemoglobin A1c% at both baseline and endline of intervention
Fasting insulin level | one year
  Fasting insulin level in µIU/mL at both baseline and endline of intervention.
Fructosamine level | one year
  fructosamine in µmol/L at both baseline and endline of intervention.
Total maternal weight gain | one year
  Total maternal weight gain during pregnancy in kilograms
Weekly weight gain | one year
  weight in kilogram will be measured weekly for all participants
Insulin Therapy | one year
  Number of participants who need insulin therapy to normalize blood sugar.
Emergency caesarean section | one year
  Number of participants who need for emergency caesarean section versus vaginal delivery.
Pregnancy-induced hypertension | one year
  Number of participants with existence of hypertension (defined as a blood pressure of at least 140/90 mmHg on two occasions).
Newborn weight | one year
  The newborn weight in grams
Newborn Length | one year
  The new born length in centimeters.
Newborn head circumference | one year
  The newborn head circumference in centimeters.
Hypoglycemic | one year
  Number of newborn babies who will suffer from hypoglycemia
Shoulder dystocia | one year
  Number of newborn babies with shoulder dystocia.

CONTACTS AND LOCATIONS:
Overall Officials: Reema F Tayyem, PhD, Study Director — University of Jordan
Locations (1):
- Sabika Allehdan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kulkarni DK. Carbohydrate counting: A practical meal-planning option for people with diabetes. Clinical Diabetes 23:120-22, 2005.
- [Background] Koivusalo SB, Rono K, Klemetti MM, Roine RP, Lindstrom J, Erkkola M, Kaaja RJ, Poyhonen-Alho M, Tiitinen A, Huvinen E, Andersson S, Laivuori H, Valkama A, Meinila J, Kautiainen H, Eriksson JG, Stach-Lempinen B. Erratum. Gestational Diabetes Mellitus Can Be Prevented by Lifestyle Intervention: The Finnish Gestational Diabetes Prevention Study (RADIEL). A Randomized Controlled Trial. Diabetes Care 2016;39:24-30. Diabetes Care. 2017 Aug;40(8):1133. doi: 10.2337/dc17-er08a. Epub 2017 Jun 14. No abstract available. PMID 28615238
- [Background] Ma WJ, Huang ZH, Huang BX, Qi BH, Zhang YJ, Xiao BX, Li YH, Chen L, Zhu HL. Intensive low-glycaemic-load dietary intervention for the management of glycaemia and serum lipids among women with gestational diabetes: a randomized control trial. Public Health Nutr. 2015 Jun;18(8):1506-13. doi: 10.1017/S1368980014001992. Epub 2014 Sep 15. PMID 25222105
- [Background] Louie JC, Markovic TP, Perera N, Foote D, Petocz P, Ross GP, Brand-Miller JC. A randomized controlled trial investigating the effects of a low-glycemic index diet on pregnancy outcomes in gestational diabetes mellitus. Diabetes Care. 2011 Nov;34(11):2341-6. doi: 10.2337/dc11-0985. Epub 2011 Sep 6. PMID 21900148
- [Background] Thomas, A. M. and Gutierrez, Y.M. (2005), American Dietetic Association guide to gestational diabetes mellitus. Chicago, IL: American Dietetic Association. Received from http://www.eatright.org/Public/ProductCatalog/ SearchableProducts/104_20728.cfm. Accessed 23 January 2016.
- [Background] Kleinwechter H, Schafer-Graf U, Buhrer C, Hoesli I, Kainer F, Kautzky-Willer A, Pawlowski B, Schunck K, Somville T, Sorger M; German Diabetes Association; German Association for Gynaecology and Obstetrics. Gestational diabetes mellitus (GDM) diagnosis, therapy and follow-up care: Practice Guideline of the German Diabetes Association(DDG) and the German Association for Gynaecologyand Obstetrics (DGGG). Exp Clin Endocrinol Diabetes. 2014 Jul;122(7):395-405. doi: 10.1055/s-0034-1366412. Epub 2014 Jul 11. No abstract available. PMID 25014091
- [Derived] Allehdan S, Basha A, Hyassat D, Nabhan M, Qasrawi H, Tayyem R. Effectiveness of carbohydrate counting and Dietary Approach to Stop Hypertension dietary intervention on managing Gestational Diabetes Mellitus among pregnant women who used metformin: A randomized controlled clinical trial. Clin Nutr. 2022 Feb;41(2):384-395. doi: 10.1016/j.clnu.2021.11.039. Epub 2021 Dec 3. PMID 34999333